CLINICAL TRIAL: NCT00401765
Title: A Phase I Study of a Chimeric Antibody Against Interleukin-6 (CNTO 328) Combined With Docetaxel in Subjects With Metastatic Hormone-Refractory Prostate Cancer
Brief Title: A Study of CNTO 328 in Patients With Metastatic Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005275; C0328T04 (Other: Centocor Ortho Biotech Services, L.L.C.)
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic neoplasm; intravenous; docetaxel; monoclonal antibody
MeSH Terms: conditions — Prostatic Neoplasms | interventions — siltuximab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1A (Docetaxel and CNTO 328) (Experimental): In cohort 1A, 75 mg/m2 docetaxel will be administered in run-in phase and 75 mg/m2 docetaxel every 3 weeks and 6 mg/kg CNTO 328 every 2 weeks will be administered in the treatment phase.
  Interventions: Drug: CNTO 328; Drug: Docetaxel
- Cohort 1B (Docetaxel and CNTO 328) (Experimental): In cohort 1B, 6 mg/kg CNTO 328 will be administered in run-in phase and 75 mg/m2 docetaxel will be administered every 3 weeks plus 6 mg/kg CNTO 328 will be administered every 2 weeks in the treatment phase.
  Interventions: Drug: CNTO 328; Drug: Docetaxel
- Cohort 2 (Docetaxel and CNTO 328) (Experimental): In cohort 2, 75 mg/m2 docetaxel will be administered in run-in phase and 75 mg/m2 docetaxel plus 9 mg/kg CNTO 328 will be administered every 3 weeks in treatment phase.
  Interventions: Drug: CNTO 328; Drug: Docetaxel
- Cohort 3 (Doctaxel and CNTO 328) (Experimental): In cohort 3, 75 mg/m2 docetaxel will be administered in the run-in phase and 75 mg/m2 docetaxel plus 12 mg/kg CNTO 328 will be administered every 3 weeks in treatment phase.
  Interventions: Drug: CNTO 328; Drug: Docetaxel

INTERVENTIONS:
Drug: CNTO 328 — Patients will receive 6 mg/kg CNTO 328 in treatment phase of cohort 1A and cohort 1B; 9 mg/kg CNTO 328 in treatment phase of cohort 2; and 12 mg/kg CNTO 328 in treatment phase of cohort 3.
Drug: Docetaxel — Patients will receive 75 mg/m2 docetaxel in run-in phase of cohort 1A, cohort 2, and cohort 3; and in treatment phase of cohort 1A, cohort 1B, cohort 2, and cohort 3.

SUMMARY:
The purpose of this study is to determine the safety of docetaxel and CNTO 328 when given together as a treatment. The second goal of this study is to determine if a combination of docetaxel and CNTO 328 has an effect on prostate cancer.

DETAILED DESCRIPTION:
This is a Phase 1 open-label, multicenter, nonrandomized study of the safety and pharmacokinetics of the combination of CNTO 328 and docetaxel in patients with metastatic Hormone-Refractory Prostate Cancer (HRPC). Eligible patients must be age >= 18 years, have histologically or cytologically confirmed adenocarcinoma of the prostate, and have documented metastatic disease. Prior chemotherapy for metastatic disease is not allowed.The study will last for approximately 26 months. This study will be conducted in 4 phases: 1. Screening (up to 4 weeks): understanding and signing an informed consent form, physical/neurological exam, an ECG, vitals will be checked, urinalysis, a radiologic assessment, routine blood samples, study blood samples, a circulating tumor cell blood sample, a testosterone level blood sample, and a prostate specific antigen (PSA) sample. If the results show that the patient can be a part of the study, the patient will begin the run-in phase. If the results of the screening show that the patient cannot be part of the study, the patient will not receive docetaxel as part of this study or CNTO 328.Starting with the first docetaxel infusion, the patient will be required to take prednisone twice a day, until the end of Cycle 3. After Cycle 3, the study doctor will decide if and/or when the prednisone taken. Dexamethasone will be required at 12 hours, 3 hours, and 1 hour before the start of every docetaxel infusion through Cycle 3. After Cycle 3, the study doctor will decide how the dexamethasone will be taken. Antiemetics (to prevent nausea and vomiting) are also required. The study doctor will decide the dose, how often, and how these should take them 2. Run-in Phase (up to 3 weeks):The term run-in phase describes a period of time before the start of the formal study treatment. During this phase, the patient will receive only one drug, either docetaxel or CNTO 328 depending on the assigned group. Groups 1A, 2, and 3: The patient will be given docetaxel 3 weeks before the formal study treatment begins. During the next 2 weeks the patient will not receive any study drug, but will undergo certain tests and procedures. Group 1B: The patient will be given a CNTO 328 infusion 2 weeks before the formal study treatment begins. During the next week the patient will not receive any study drug, but will have certain tests and procedures. 3. Cycles 1 through 17 (14 cycles - up to 46 weeks and with additional 3 cycles -up to 55 weeks):Cycles 1 through 17 are each planned to be 3 weeks in length. All treatment groups will receive an infusion of docetaxel on week 1 of every cycle. The CNTO 328 infusion occurs based on the treatment group to which the patients are assigned. Group 1A: Patients will receive a 6mg/kg infusion of CNTO 328 every two weeks, starting on week 1, cycle 1. Group 1B: Patients will receive a 6mg/kg infusion of CNTO 328 every two weeks, starting two weeks prior to cycle 1.Group 2: Patients will receive a 9 mg/kg infusion of CNTO 328 every three weeks, starting on week 1, cycle 1. Group 3: Patients will receive a 12mg/kg infusion of CNTO 328 every three weeks, starting on week 1, cycle 1. The overall amount of CNTO 328 increases with each higher group. Therefore, Group 1A and 1B will be filled before Group 2, and Group 2 will be filled before Group 3. This allows CNTO 328 to be tested in a safer manner. The docetaxel dose remains the same for all three groups.Patients may receive up to 14 cycles of treatment provided there is no evidence of disease progression, including serum PSA progression, or unacceptable toxicity. However, patients responding to treatment with at least stable disease (SD) after 14 cycles will be permitted to receive 3 additional cycles of treatment. In addition to drug therapy, patients will receive other tests and procedures. Most of the tests required before study medication is administered and throughout the study would be done normally during any treatment for prostate cancer. However, these tests and procedures may be done more often. The following are the tests and procedures: Routine blood tests; Study blood samples; Testosterone level sample; PSA sample; Circulating Tumor Cell blood sample; Urinalysis; Physical exam/neurological exam; Vital signs; ECG (electrocardiogram); Radiological tests4. Follow-up: After patients complete treatment they will have follow-up visits including patients that discontinue treatment early. The patients will have them 1, 2, 3, and 4 weeks after the final treatment cycle is completed. The Week 4 visit will be the "End of Study Visit". There will be 3 more visits at 12, 18, and 24 weeks after the final treatment cycle. Long-term Follow-up: No matter when or why the patients leave the study, the study doctor or nurse may telephone them to ask about their health and/or look at their medical records every 3 months to check on how they are doing. They will do this for one year after the last infusion of study drug. Patients will not need to go to the study center or have any tests performed. The study center will also ask about any treatment the patient received after they completed their participation in the study . Docetaxel 75 mg/m2 will be given intravenously (into the vein) once every 3 wks for up to 17 three week cycles. CNTO328 will be administered intravenously (into the vein) over 2 hours according to one of the following regimens: 6 milligrams of medication per kilogram of body weight (mg/kg) once every 2 wks; 9 mg/kg once every 3 wks; and 12 mg/kg every 3 wks for up to 17 three week cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Radiologically documented metastatic disease
* No prior systemic chemotherapy for metastatic hormone refractory prostate cancer
* Progressive hormone-refractory disease after orchiectomy or gonadotropin-releasing hormone analog and/or anti-androgen treatment within 12 months of screening based on 1 of the following: Transaxial imaging tumor progression, Rise in 2 consecutive prostate-specifec antigen (PSA) values obtained at least 7 days apart or Radionucleotide bone scan progression
* Karnofsky performance status of greater than or equal to 60

Exclusion Criteria:

* Prostate cancer that does not express serum PSA or is less than 5.0 ng/mL at screening
* Received any investigational drug/agent within 30 days or 5 half-lives, whichever is longer
* Prior malignancy (other than prostate cancer) except adequately treated basal cell or squamous cell carcinoma of the skin or other cancer for which the subject has been disease-free for greater than or equal to 3 years
* Known central nervous system metastases
* Received any over-the-counter or herbal treatment for prostate cancer (eg, PC SPES [an herbal refined powder]) within 4 weeks prior to screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Number of Patients With Adverse Events as a Measure of Safety and Tolerability | Up to 1 year after the last study medication administration
Plasma Concentration of Docetaxel | predose, post dose (up to 6 hours), and Week 4 (end of treatment visit)
Serum Concentration of Docetaxel in Combination With CNTO 328 | predose, post dose (up to 6 hours), and up to Week 4 (end of treatment visit)

SECONDARY OUTCOMES:
Number of Patients with Prostate-Specific Antigen (PSA) Response | Screening phase (within 4 weeks before administration), every 3 weeks up to 14 cycles or progressive disease, whichever comes first
  PSA response is defined as number of patients with 50% or more reduction in serum PSA below the baseline value.
Number of Patients With PSA Reduced Within 3 Months | Screening phase (within 4 weeks before administration), every 3 weeks up to 14 cycles or progressive disease, whichever comes first
  PSA reduced within 3 months is defined as number of patients with 50% or more reduction in serum PSA below the screening value within 3 months after the first administration of study medication.
PSA Progression in Patients | Screening phase (within 4 weeks before administration), every 3 weeks up to 14 cycles or progressive disease, whichever comes first
Duration of Tumor Response | Screening phase (within 4 weeks before administration); every 3 weeks up to 14 cycles; and every 3 months up to 1 year after the last study medication administration
  Duration of tumor response is defines as the time from first documented evidence of response (complete response [Total disappearance of a disease] or partial response [50% or more decrease from baseline in the sum of products of perpendicular diameters of all measurable lesions]) to documented disease progression or death, whichever is earlier.
Duration of PSA response | Screening phase (within 4 weeks before administration), every 3 weeks up to 14 cycles or progressive disease, whichever comes first
  Duration of PSA response is defined as the time from first observation of serum PSA response until PSA progression, disease progression, or death, if sooner.
Objective Tumor Response | Screening phase (within 4 weeks before administration); every 3 weeks up to 14 cycles; and every 3 months up to 1 year after the last study medication administration
  Tumor response will be evaluated as Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD). CR is defined as complete disappearance of all measurable and evaluable disease; PR is defined as 50 percentage or more decrease from baseline in the sum of products of diameters of all measurable lesions; SD is defined as 25 percentage or less decrease from baseline in the sum of products of diameters of all measurable lesions; and PD is defined as 25 percentage or more increase in the sum of products of diameters of measurable lesions over the smallest sum observed, or reappearance of any lesion which had disappeared, or appearance of any new lesion, or failure to return for evaluation due to death or deteriorating condition.
Pharmacodynamics of CNTO 328 administered in combination with docetaxel | predose, post dose (up to Day 14), and up to Week 4 (end of treatment visit)
  Pharmacodymanics parameters: C reactive protein, Interleukin-6 (IL-6), serum amyloid-A, serum prostate-specific antigen, IL-6 bioactivity, vascular endothelial growth factor, fibroblast growth factor, and circulating tumor cells will be measured.
Serum concentration of CNTO 328 | predose, post dose (up to Day 14), and up to Week 4 (end of treatment visit)
Serum concentration of CNTO 328 in combination with docetaxel | predose, post dose (up to Day 14), and up to Week 4 (end of treatment visit)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (5):
- United States (5):
  - Baltimore, Maryland
  - New York, New York
  - Chapel Hill, North Carolina
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee

REFERENCES:
- See also: A Phase 1 Study of a Chimeric Antibody Against Interleukin-6 (CNTO 328) Combined with Docetaxel in Subjects with Metastatic Hormone-Refractory Prostate Cancer — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=158&filename=CR005275_CSR.pdf